CLINICAL TRIAL: NCT05932459
Title: A Phase I Clinical Study to Evaluate the Bioavailability, Food Effect and Pharmacokinetic Characteristics of Oral Deuremidevir Hydrobromide for Suspension in Chinese Healthy Volunteers
Brief Title: A Study to Evaluate the Bioavailability, Food Effect and Pharmacokinetics of Deuremidevir Hydrobromide for Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VV116-RSV-01
Record Dates: First submitted 2023-06-21; First posted 2023-07-06 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2023-06

CONDITIONS: Healthy Subjects
Keywords: VV116-RSV; Bioavailability; Food effect; Pharmacokinetics
MeSH Terms: interventions — Suspensions; GS-621763

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- BA Study (Experimental): 18 subjects were randomly divided into two sequences, TR and RT, with 9 subjects in each sequence, and were given in fasted condition once per period. In the first period of TR sequence, 100mg Deuremidevir Hydrobromide dry suspension was taken, and in the second period, 100 mg Deuremidevir Hydrobromide tablets were taken. In the first period of RT sequence, 100mg Deuremidevir Hydrobromide tablets were taken, and 100mg Deuremidevir Hydrobromide dry suspension was taken in the second period.
  Interventions: Drug: Deuremidevir Hydrobromide for Suspension 100mg; Drug: Deuremidevir Hydrobromide tablets 100mg
- FE Study (Experimental): 12 subjects were randomly divided into two sequences, sequence 1 and sequence 2. There were 6 subjects in each sequence, and one dose per period. Sequence 1: Take Deuremidevir Hydrobromide dry suspension in fasted condition in period 1, and take Deuremidevir Hydrobromide dry suspension after taking infant formula for 10 minutes in period 2; Sequence 2: Take Deuremidevir Hydrobromide dry suspension after taking infant formula for 10 minutes in period 1, and take Deuremidevir Hydrobromide dry suspension in fasted condition in period 2.
  Interventions: Drug: Deuremidevir Hydrobromide for Suspension 300mg
- PK Study (Experimental): Fasting; PK study form is dry suspension, the doses are 25 mg, 100 mg, 300 mg, taken orally once in fasted condition. 8 subjects in 25 mg group; The 100 mg group used the data of 18 subjects with dry suspension in BA study, while the 300 mg group used the fasting condition data of 12 subjects with dry suspension in FE study.
  Interventions: Drug: Deuremidevir Hydrobromide for Suspension 100mg; Drug: Deuremidevir Hydrobromide for Suspension 300mg; Drug: Deuremidevir Hydrobromide for Suspension 25mg

INTERVENTIONS:
Drug: Deuremidevir Hydrobromide for Suspension 100mg — Take it with 240ml water in fasted condition.
  Other Names: VV116
  Arms: BA Study; PK Study
Drug: Deuremidevir Hydrobromide for Suspension 300mg — Take it with water in fasted condition or after taking infant formula.
  Other Names: VV116
  Arms: FE Study; PK Study
Drug: Deuremidevir Hydrobromide for Suspension 25mg — Take it with 240ml water on an empty stomach.
  Other Names: VV116
  Arms: PK Study
Drug: Deuremidevir Hydrobromide tablets 100mg — Take it with 240ml water in fasted condition.
  Other Names: VV116
  Arms: BA Study

SUMMARY:
This study is divided into three parts: bioavailability study (hereinafter referred to as "BA study"), food effect study (hereinafter referred to as "FE study") and pharmacokinetic characteristics study (hereinafter referred to as "PK characteristics study"). A total of 38 subjects are planned to be enrolled. The three parts of the study can be carried out simultaneously, and there is no order requirement. The subjects will be assigned to one of them according to the enrollment order. Dose selection is 100mg, 300mg and 25mg.

DETAILED DESCRIPTION:
BA study plan included 18 subjects, in the form of dry suspension and tablets, with a dose of 100 mg. Subjects were randomly divided into two sequences, TR and RT, with 9 cases in each sequence. They were given once in fasted condition each period, and the dry suspension and tablets were designed in a double crossover way.

12 subjects were enrolled in the FE study plan, and the dose was 300mg in dry suspension. Subjects were randomly divided into two sequences, sequence 1 and sequence 2, with 6 cases in each sequence, and given once per period. Fasting and infant formula milk double crossover were tested in two periods according to the administration sequence.

PK study form is dry suspension, the doses are 25 mg, 100 mg, 300 mg, taken orally once in fasted condition. 8 subjects will be enrolled in the 25mg group. The 100 mg group used the data of 18 subjects with dry suspension in BA study, while the 300 mg group used the fasting condition data of 12 subjects with dry suspension in FE study. The 100 mg and 300 mg groups will not be enrolled separately.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 60 years old, males or females;
2. Body weight no less than 40 kg, Body Mass Index of 18.5 to 27.0kg/m2;
3. Vital signs examination, physical examination, laboratory examination and electrocardiogram examination results were normal or abnormal without clinical significance;
4. Subjects who are willing to take proper contraceptive during the study and within 3 months after the study completed;
5. Subjects who are able to understand and follow study plans and instructions; Subjects who have voluntarily decided to participate in this study, and signed the informed consent form.

Exclusion Criteria:

1. Subjects with hypersensitivity to deuremidevir hydrobromide for suspension or any of the excipients;
2. Subjects with allergic diseases or allergic constitution;
3. Subjects who are allergic to formula ingredients or lactose intolerant or unable to ingest infant formula (only applicable to FE research);
4. Subjects with central nervous system, cardiovascular system, gastrointestinal, respiratory system, urinary, Hematologic System, metabolic disorders that require medical intervention or other diseases (such as psychiatric history) that are not suitable for clinical trials;
5. Subjects with acute upper respiratory tract infection within 2 weeks before screening;
6. Subjects who have received blood transfusion or used blood products within 3 months before screening or who have lost more than ≥400 mL of blood due to other reasons (except female physiological blood loss);
7. Subjects who have participated in clinical trials of other drugs within 3 months before screening;
8. Subjects who have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines or health products orally within 2 weeks before screening;
9. Being a drug addict or alcohol addict within one year before screening, being an alcoholic at present or in the past (drinking more than 14 standard units per week, and one standard unit contains 14 g of alcohol, such as 360 mL of beer or 45 mL of strong liquor with 40% alcohol content or 150 mL of wine), or being positive in alcohol breath test;
10. Subjects who smoked more than 5 cigarettes a day within one year before screening;
11. Subjects who can't quit smoking and drinking during the experiment;
12. Subjects who are positive for hepatitis B virus surface antigen, hepatitis C virus antibody, Treponema pallidum antibody (TPPA) or human immunodeficiency virus antibody (Anti-HIV);
13. Abnormal chest X-ray results with clinical significance;
14. Total bilirubin (TBIL) at screening or baseline > upper limit of normal value (ULN); Alanine transaminase (ALT) or aspartate transaminase (AST) > 1.5 times ULN；;
15. The glomerular filtration rate (EGFR) at screening or baseline is less than 90 ml/min;
16. Abnormal ECG at screening or baseline, single examination of QTcF (after heart rate correction) is >450 ms for male and > 470 ms for female, and/or other abnormalities with clinical significance;
17. Pregnant or lactating woman or male subjects whose spouse has a child care plan within 3 months;
18. The investigator believes that there are other factors that are not suitable for participating in this trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-07-09 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Cmax | 48 hours after administration
  maximum observed plasma concentration
AUC0-t | 48 hours after administration
  area under the plasma concentration time curve from time zero to the last measurable concentration
AUC0-∞ | 48 hours after administration
  area under the plasma concentration-time curve from time zero to infinity
AUC0-24h | 48 hours after administration
  Area under the plasma concentration-time curve from 0 to 24 hours
Tmax | 48 hours after administration
  time at which Cmax occurs
Tlag | 48 hours after administration
  time lag
t1/2z | 48 hours after administration
  half life of elimination
CLz/F | 48 hours after administration
  apparent clearance
Vz/F | 48 hours after administration
  apparent volume of distribution during the terminal phase

SECONDARY OUTCOMES:
AE & SAE | From Day1 to Day10 after administration
  Adverse event & serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, Principal Investigator — Hushan Hospital of the Fudan university; Xiaojie Wu, Principal Investigator — Hushan Hospital of the Fudan university
Locations (1):
- Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No